CLINICAL TRIAL: NCT02680366
Title: A Multi-center, Randomized, Single-blind, Controlled Clinical Trial of Treatment of Severe Asherman Syndrome by Collagen Scaffold Loaded With Autologous Bone Marrow Mononuclear Cells
Brief Title: Treatment of Severe Asherman Syndrome by Collagen Scaffold Loaded With Autologous Bone Marrow Mononuclear Cells
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: Changzhou Maternal and Child Care Hospital (Other)
Responsible Party: Principal Investigator, Yali Hu, MD,PhD, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201600301
Record Dates: First submitted 2016-01-30; First posted 2016-02-11 (Estimated); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Infertility; Asherman Syndrome
MeSH Terms: conditions — Infertility; Gynatresia

STUDY DESIGN:
Intervention Model Description: BMSCs group (BMSCs-scaffold plus Foley catheter) or control group (only Foley catheter).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- collagen/ABMNC scaffold (Experimental): collagen/ABMNC scaffold covered on Foley catheter balloon inserted after hysteroscopic adhesiolysis
  Interventions: Device: collagen/ABMNC scaffold
- Foley catheter balloon (Active Comparator): Foley catheter balloon inserted after hysteroscopic adhesiolysis
  Interventions: Device: Foley catheter balloon

INTERVENTIONS:
Device: collagen/ABMNC scaffold — The patients will receive a bone marrow puncture to collect bone marrow cells which are used to isolation of ABMNCs. After that, hysteroscopic adhesiolysis will be done according to the patient's uterine adhesion. Then, the collagen/ABMNCs scaffold was covered on a Foley catheter balloon and placed into the uterine cavity. The catheter balloon was kept for 24 hours and then removed. Oral antibiotics were given to prevent infection in the second and third days after operation. 72 hours after the surgery, a vaginal speculum examinations will be done in order to make patients unknown about their arms. Estrogen will be administrated for 3 cycles to support the endometrial regeneration after the surgery. The clinical follow up will be done at 1, 3 and 6 months after the procedure.
  Arms: collagen/ABMNC scaffold
Device: Foley catheter balloon — The patients will receive a sham bone marrow puncture which just has a local anesthesia and collects no bone marrow cells to isolation. After that, hysteroscopic adhesiolysis will be done according to the patient's uterine adhesion. And then, a Foley catheter balloon will be placed into the uterine cavity and kept for 72 hours before it is removed. Oral antibiotics were given to prevent infection in the second and third days after operation. Estrogen will be administrated for 3 cycles to support the endometrial regeneration after the surgery. The clinical follow up will be done at 1, 3 and 6 months after the procedure.
  Arms: Foley catheter balloon

SUMMARY:
This study evaluates the addition of collagen scaffold loaded with autologous bone marrow mononuclear cells(ABMNC) to Foley catheter balloon after hysteroscopic adhesiolysis in the treatment of severe asherman syndrome. Half of participants will receive collagen/ABMNC scaffold after hysteroscopic adhesiolysis, while the other half will receive Foley catheter balloon.

DETAILED DESCRIPTION:
Severe asherman syndrome will lead to infertility, and the most common method to treat asherman syndrome is operating to dissect adhesions. In order to prevent the postoperative re-adhesion, many physical isolation measures have been tried. However, they don't improve the microenvironment of endometrial regeneration. It's reported that bone marrow mononuclear cells have good effects on the functional recovery of injured uterus. This study will determine whether collagen scaffolds loaded with autologous bone marrow mononuclear cells will be more effective than Foley balloon catheters at treating infertile women with severe intrauterine adhesions who have taken hysteroscopic adhesiolysis. In addition, the study will be carried out in 2 centers, one is the Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, the other is Changzhou Maternal and Child Health Care Hospital that is in Jiangsu Province.

ELIGIBILITY:
Inclusion Criteria:

* Having a clear desire to fertility;
* Infertility that is defined as a women fails to become pregnant after having a normal sex life for two years without contraception.
* Hysteroscopy examination confirmed intrauterine adhesions(patients who has at least one of the three symptoms which are amenorrhea, hypomenorrhea or infertility, and hysteroscopy or histologic diagnosis of intrauterine adhesions), meeting American Fertility Society diagnostic criteria Ⅱ-III;
* Normal ovarian function;
* Regular Menstrual cycles and menstruation is normal before abortion or curettage;
* BMI< 30 kg/m2;
* Sign a consent form;
* Follow the test plan and follow-up process.

Exclusion Criteria:

* Hereditary diseases;
* Simple thin endometrium with no uterine cavity adhesion;
* Simple Uterine scar formation with no uterine cavity adhesion after hysteroscopic adhesiolysis;
* Contraindications to bone marrow collection or assisted reproductive technology;
* History of malignant tumor;
* Other diseases associated with the uterus: uterine fibroids, severe adenomyosis, severe malformations of the uterus;
* Abnormal blood coagulation, liver and kidney dysfunction, or other diseases which the researchers think may affect the study(such as: uncontrolled hypertension, diabetes, sexually transmitted diseases);
* With a positive urine pregnancy test；
* Participating in other clinical studies at the same time;
* Hysteroscopic adhesiolysis more than 3 times in the past.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 152 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | up to 24 months
  A successful clinical pregnancy means that at the 12th week of pregnancy, ultrasound reveals that the fetus had a heart activity and the size of the fetus is in consistent with the gestational week.

SECONDARY OUTCOMES:
Menstrual volumes and menstrual improvement: | at 3 and 6 months post-operation
  PBAC scores in the third and sixth menstrual cycles after the initial adhesiolysis and PBAC scores increase compared to pre-operation
Maximal endometrial thickness | at 3 and 6 months post-operation
  Measure the endometrial thickness during ovulation by ultrasound by the same trained medical sonographers at 3 and 6 months after surgery, comparing with pre-operation.
Re-adhesion rate at the second-look hysteroscopy | at 3 months post-operation
AFS score at the second-look hysteroscopy and AFS score decrease compared to pre-operation | at 3 months post-operation
Miscarriage rate | up to 24 months
preterm birth rate | up to 24 months
ectopic pregnancy rate | up to 24 months
live birth rate | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Yali Hu, MD,PhD, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Both the study protocol and the statistical analysis plan are available on request.
Supporting Information: Study Protocol, SAP
Time Frame: The data are available on reasonable request beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal will be given access to the data to achieve aims in the proposal.